CLINICAL TRIAL: NCT03684590
Title: A Prospective, Randomized, PACU Blinded Study to Compare ANI-guided Analgesic Administration Versus Standard Care in Surgical Patients Receiving Balanced Sevoflurane-Fentanyl Anesthesia
Brief Title: ANI Versus Standard Care in Surgical Patients Receiving Balanced Sevoflurane-Fentanyl Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2018-0096
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard opioid administration (Active Comparator): Intraoperative opioid will be administered by guiding standard practice
  Interventions: Other: Standard opioid administration
- ANI-guided opioid administration (Experimental): Intraoperative opioid will be administered based on the analgesia nociceptive index (ANI)
  Interventions: Device: ANI-guided opioid administration

INTERVENTIONS:
Device: ANI-guided opioid administration — Intraoperative opioid will be administered guided by analgesia nociceptive index (ANI) values measured by ANI monitor (MetroDoloris Medical Systems, Lille, France)
  Arms: ANI-guided opioid administration
Other: Standard opioid administration — Intraoperative opioid will be administered according to standard practice during surgery.
  Arms: Standard opioid administration

SUMMARY:
This study aims to be a randomized, controlled study of ANI-guided opioid administration versus standard clinical practice in surgical patients undergoing general anesthesia with balanced sevoflurane-fentanyl. Patients will be randomly assigned to 2 groups- ANI vs. standard care. The intraoperative and postoperative management of all patients will be standardized by protocol. The PACU nurses and postop assessor will be blinded as to which group the patient is in.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* ASA 1-2
* BMI 19-35 kg/m2
* Patients undergoing surgery with general anesthesia with sevoflurane- fentanyl
* Planned abdominal or spinal surgery lasting 1-3 hours
* Willing and able to consent in English or Spanish
* No current history of advanced pulmonary or cardiovascular disease

Exclusion Criteria:

* Age less than 18 or older than 75
* Patient does not speak English or Spanish
* Patient refusal
* Monitored anesthesia care (MAC) or regional anesthesia planned
* Pregnant or nursing women
* "Stat" (emergent) cases
* ECG rhythm other than regular sinus rhythm
* Implanted pacemakers
* On antimuscarinic agents, alpha 2 agonists, antiarrhythmics, or beta blockers
* Presence of pacemaker
* Autonomic nervous system disorder
* Use of chronic opioids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Boselli E, Daniela-Ionescu M, Begou G, Bouvet L, Dabouz R, Magnin C, Allaouchiche B. Prospective observational study of the non-invasive assessment of immediate postoperative pain using the analgesia/nociception index (ANI). Br J Anaesth. 2013 Sep;111(3):453-9. doi: 10.1093/bja/aet110. Epub 2013 Apr 16. PMID 23592690
- [Background] Bluth T, Pelosi P, de Abreu MG. The obese patient undergoing nonbariatric surgery. Curr Opin Anaesthesiol. 2016 Jun;29(3):421-9. doi: 10.1097/ACO.0000000000000337. PMID 26982116
- [Background] Budiansky AS, Margarson MP, Eipe N. Acute pain management in morbid obesity - an evidence based clinical update. Surg Obes Relat Dis. 2017 Mar;13(3):523-532. doi: 10.1016/j.soard.2016.09.013. Epub 2016 Sep 19. PMID 27771314
- [Background] Lovich-Sapola J, Smith CE, Brandt CP. Postoperative pain control. Surg Clin North Am. 2015 Apr;95(2):301-18. doi: 10.1016/j.suc.2014.10.002. Epub 2015 Jan 24. PMID 25814108
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Borsook D, Kussman BD, George E, Becerra LR, Burke DW. Surgically induced neuropathic pain: understanding the perioperative process. Ann Surg. 2013 Mar;257(3):403-12. doi: 10.1097/SLA.0b013e3182701a7b. PMID 23059501
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Jeanne M, Clement C, De Jonckheere J, Logier R, Tavernier B. Variations of the analgesia nociception index during general anaesthesia for laparoscopic abdominal surgery. J Clin Monit Comput. 2012 Aug;26(4):289-94. doi: 10.1007/s10877-012-9354-0. Epub 2012 Mar 28. PMID 22454275
- [Background] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Background] Sabourdin N, Arnaout M, Louvet N, Guye ML, Piana F, Constant I. Pain monitoring in anesthetized children: first assessment of skin conductance and analgesia-nociception index at different infusion rates of remifentanil. Paediatr Anaesth. 2013 Feb;23(2):149-55. doi: 10.1111/pan.12071. Epub 2012 Nov 21. PMID 23170802
- [Background] Upton HD, Ludbrook GL, Wing A, Sleigh JW. Intraoperative "Analgesia Nociception Index"-Guided Fentanyl Administration During Sevoflurane Anesthesia in Lumbar Discectomy and Laminectomy: A Randomized Clinical Trial. Anesth Analg. 2017 Jul;125(1):81-90. doi: 10.1213/ANE.0000000000001984. PMID 28598927
- [Background] Szental JA, Webb A, Weeraratne C, Campbell A, Sivakumar H, Leong S. Postoperative pain after laparoscopic cholecystectomy is not reduced by intraoperative analgesia guided by analgesia nociception index (ANI(R)) monitoring: a randomized clinical trial. Br J Anaesth. 2015 Apr;114(4):640-5. doi: 10.1093/bja/aeu411. Epub 2014 Dec 23. PMID 25540069
- [Background] Dundar N, Kus A, Gurkan Y, Toker K, Solak M. Analgesia nociception index (ani) monitoring in patients with thoracic paravertebral block: a randomized controlled study. J Clin Monit Comput. 2018 Jun;32(3):481-486. doi: 10.1007/s10877-017-0036-9. Epub 2017 Jun 19. PMID 28631050

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Opioid Administration | ANI-guided Opioid Administration
Started | 49 | 53
Completed | 49 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Opioid Administration | ANI-guided Opioid Administration | Total
Number analyzed (Participants) | 49 | 53 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 52 | 101
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 42.69 [23 to 61] | 45.31 [29 to 67] | 43.87 [23 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 52 | 101
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 37 | 68
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 53 | 102

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Severe Postoperative Pain
Description: The primary outcome will be the NRS pain scores reported during recovery
Time Frame: postoperative recovery period, an average of 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Opioid Administration | ANI-guided Opioid Administration
Number analyzed (Participants) | 49 | 53
Participants | 49 | 53

2. Secondary Outcome: The Incidence of Pain Medication Use
Description: The total amounts of opioid analgesics administered in the operating room (OR) and post-anesthesia care unit (PACU)
Time Frame: Perioperative and postoperative recovery period
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Standard Opioid Administration | ANI-guided Opioid Administration
Number analyzed (Participants) | 49 | 53
micrograms | 224.1 (140.5) | 294.4 (170.3)

3. Secondary Outcome: The Incidence of Postoperative Nausea/Vomiting in Post-anesthesia Care Unit (PACU)
Description: The incidence of nausea/vomiting reported during recovery
Time Frame: Postoperative recovery period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Opioid Administration | ANI-guided Opioid Administration
Number analyzed (Participants) | 49 | 53
Participants | 0 | 0

4. Secondary Outcome: The Incidence of Minimal Pain
Description: The percent of subjects with minimal pain (NPS < 3) in post-anesthesia care unit (PACU)
Time Frame: Postoperative recovery period
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Opioid Administration | ANI-guided Opioid Administration
Number analyzed (Participants) | 49 | 53
Participants | 12 | 22

ADVERSE EVENTS:
Time Frame: 24 hours post-op
Description: All patients that were enrolled were healthy individuals and therefore not at risk for adverse events.
Arm/Group | Standard Opioid Administration | ANI-guided Opioid Administration
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/53
Other Adverse Events (participants affected / at risk) | 0/49 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03684590/Prot_SAP_000.pdf